CLINICAL TRIAL: NCT03124303
Title: Interventions for Postoperative Delirium: Biomarker-3
Acronym: IPOD-B3
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2015-0374; 1K23AG055700-01A1 (NIH); 1R01AG063849-01 (NIH); A530900 (Other: UW Madison); SMPH\ANESTHESIOLOGY (Other: UW Madison); Protocol Version 1/15/25 (Other: UW Madison)
Record Dates: First submitted 2017-03-29; First posted 2017-04-21 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium | interventions — Magnetic Resonance Spectroscopy; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participant blood and cerebrospinal fluid (CSF) will be collected and stored for future analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Participants 1-320: First 320 participants enrolled
  Interventions: Procedure: High Density-Electroencephalogram; Procedure: Magnetic Resonance Imaging
- Participants 321-470: Final 150 participants enrolled
  Interventions: Procedure: High Density-Electroencephalogram; Procedure: Magnetic Resonance Imaging; Procedure: Blood specimen collection; Diagnostic Test: Pupillometry

INTERVENTIONS:
Procedure: High Density-Electroencephalogram — EEG is a safe non-invasive technology without complications that may be used to help diagnose delirium
  Other Names: EEG
Procedure: Magnetic Resonance Imaging — MRI scan of brain
  Other Names: MRI
Procedure: Blood specimen collection — Blood will be collected from participants
  Groups: Participants 321-470
Diagnostic Test: Pupillometry — A pupillometer is a device that measures the size of the pupils.
  Groups: Participants 321-470

SUMMARY:
The IPOD-B3 study aims to characterize the relationship between premorbid brain activity and postoperative delirium in patients undergoing major surgery. This is a expansion of the NeuroVISION Bolt-On study, NCT01980511.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1: Age ≥65 years
* Cohort 2: Age ≥60 years
* Anticipated length of hospital stay of at least 2 days after surgery that occurs under general or neuraxial anesthesia
* Written Informed Consent for potential participation prior to surgery

Exclusion Criteria:

* Contraindication to EEG
* Unable or unwilling to attend the follow-up appointments
* Documented history of dementia
* Deemed incapable of providing consent by surgical team
* Residing in a nursing home
* Undergoing intracranial surgery
* Unable to complete neurocognitive testing due to language, vision or hearing impairment
* Unable to communicate with the research staff due to language barriers
* For optional MRI portion of the study: Contraindication to MRI (e.g., implanted devices not safe for MRI studies, claustrophobia, unable to lie flat or still)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort 1: Patients, 65 years of age and older, undergoing surgery with an estimated length of stay of 2 days or greater.
  Cohort 2: Patients, 60 years of age and older, undergoing surgery with an estimated length of stay of 2 days or greater.
Sampling Method: Non-Probability Sample
Enrollment: 468 (Estimated)
Dates: Start 2017-02-13 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Functional Connectivity | Pre-operative measure: Up to 4 weeks prior to surgery. Post-operative measure: Post-Operative days 1-4
  Change from baseline functional connectivity at immediate postoperative period and association between delirium (CAM) and functional connectivity of the cingulate cortex
Brain state change | Post-operative day 1 through 4
  Quantified by the MSD across regions of interest from resting state time-series to randomly spaced points across the time-series. Measured for Cohort 2 only.

SECONDARY OUTCOMES:
Inflammation | Pre-operative measure: Up to 4 weeks prior to surgery. Post-operative measure: POD1-4
  Assess the changes from preoperative to postoperative EEG associated with delirium and change in plasma/cerebrospinal fluid (CSF) IL-6 or other biomarkers (e.g. other cytokines or markers of neronal injury)
Biomarkers | Post-operative day 1 through 4
  Identify biomarkers of delirium and neural damage through changes in circulating plasma proteins and molecules (through mass spectometry)
Brain measurements | Preoperative MRI will occur up to 4-weeks prior to surgery. Delirium is followed postoperatively, days 1-4
  Assess the association between preoperative white matter connectivity (DTI) and cortical thickness (derived from MRI) and postoperative delirium
Long term cognition | Pre-operative cognition measures will occur up to 4 weeks prior to surgery. Post-operative delirium measured on postoperative days 1-4. Long term post-operative cognition measured 1 year after surgery.
  Examine the incidence of delirium with change in cognition from preoperatively to one-year postoperatively.
Long term cognition | Pre-operative measure: Up to 4 weeks prior to surgery. Post-operative measure: Up to two years after surgery
  Assess the impact of delirium, preoperative and postoperative imaging biomarkers with a change in long term cognition
Baseline cognition, specific and global. | Cognition is assessed preoperatively. Participants are followed for delirium on postoperative days 1-4
  Examine the association between preoperative cognition using a neuropsychological battery, and postoperative delirium incidence.
Biomarkers and brain measurements | Pre-op measures: up to 4 weeks prior to surgery. Post-op measures: one year, and two years, after surgery.
  Assess the changes in cognition and biomarkers over one year with EEG changes.
Representativeness of surgical population | Pre-op MRI: up to 4 weeks prior to surgery.
  Identify whether patients who consent to the MRI are reflective of the surgical population.
Genetics and delirium | Pre-op blood collected up to 4 weeks prior to surgery. Post-operative delirium measured on postoperative days 1-4. Post-operative blood collected on postoperative days 1-4. Long term blood collected 90 days and 1 year after surgery.
  Identify genetic and epigenetic changes associated with delirium and its pathogenesis.
Postoperative amyloid beta deposition and delirium | Post-operative delirium measured on postoperative days 1-4. PET imaging will occur 90 days after surgery.
  Identify associations between delirium and amyloid beta deposition detected by Positron Emission Tomography at 90 days after surgery in sub-study IPOD-PET.
Long term changes in amyloid beta deposition and delirium | Pre-operative PET imaging will occur up to 4 weeks prior to surgery. Post-operative delirium measured on postoperative days 1-4. Post-operative PET imaging will occur 1 year after surgery.
  Identify associations between delirium and amyloid beta deposition detected by Positron Emission Tomography preoperatively and 1 year after surgery in sub-study IPOD-PET2.
Long term cognition | Pre-operative cognition measures will occur up to 4 weeks prior to surgery. Long term post-operative cognition measured 2 years after surgery.
  Identify predictors of delirium severity and incidence, for change in cognition from preoperatively to two-years postoperatively.
Mismatch negativity | Post-operative day 1 through 4
  EEG mismatch negativity during delirium compared to resolution of delirium.
Resolution of slow wave activity | Post-operative day 1 through 4
  Slow wave activity during delirium compared to resolution of delirium.
Connectivity during delirium | Post-operative day 1 through 4
  Dynamic causal modeling of cortical connectivity during delirium.
Effects of inflammation on brain activity | Post-operative day 1 through 4
  EEG correlations with biomarkers of inflammation and neuronal injury.
Delirium subtypes - neuronal dynamics | Post-operative day 1 through 4
  EEG neuronal dynamics (energy landscape analysis) during hyperactive vs hypoactive delirium.
Delirium subtypes - predisposing neuronal dynamics | Up to 4 weeks prior to surgery.
  Preoperative neuronal dynamics between hyperactive and hypoactive delirium.
Delirium subtypes - network stitching | Post-operative day 1 through 4
  Task evoked network switching and locus coeruleus activity between hyperactive and hypoactive delirium.
Delirium subtypes - network integration | Up to 4 weeks prior to surgery.
  Preoperative brain network integration vs differentiation between hyperactive and hypoactive delirium.
Pupillary responses | Post-operative day 1 through 4
  Pupillary response during rest and cognitive task in delirious versus nondelirious participants.
Metabolism and SWA | Post-operative day 1 through 4
  Correlation between SWA location, delirium subtype, and MCT2 expression.
Injury versus inflammation | 4 weeks prior to surgery to 1 year post-surgery
  Delayed resolution of biomarkers of neuronal dysfunction and inflammation as competing theories to neuronal injury.
Neuronal injury - surgery type | Post-operative day 1 through 4
  Association between biomarkers of neuronal injury and type of surgery.
Change in cognition | Baseline to 1 year post-surgery
  Association of biomarkers of neuronal injury with change in cognition at 1 year.
Change in cognition | Post-operative day 1 through 4
  Association of biomarkers of neuronal injury with change in cognition.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Pearce, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taylor NL, Wehrman J, Banks MI, Nair V, Pearce RA, Kunkel D, Shine JM, Prabhakaran V, Lennertz R, Sanders RD. Dysfunctional resting state network connectivity predicts postoperative delirium after major surgery. Br J Anaesth. 2025 Dec 30:S0007-0912(25)00844-X. doi: 10.1016/j.bja.2025.11.036. Online ahead of print. PMID 41475933
- [Derived] Rivera C, Kunkel D, Her M, Qureshi S, Pearce RA, Sanders RD, Lennertz R. The 3-Minute Diagnostic Confusion Assessment Method severity score correlates with the Delirium Rating Scale-Revised-98 and with biomarkers of delirium. BJA Open. 2025 Apr 21;14:100398. doi: 10.1016/j.bjao.2025.100398. eCollection 2025 Jun. PMID 40331035
- [Derived] Kunkel D, Parker M, Casey C, Krause B, Taylor J, Pearce RA, Lennertz R, Sanders RD. Impact of perioperative inflammation on days alive and at home after surgery. BJA Open. 2022 Apr 14;2:100006. doi: 10.1016/j.bjao.2022.100006. eCollection 2022 Jun. PMID 37588271
- [Derived] Taylor J, Wu JG, Kunkel D, Parker M, Rivera C, Casey C, Naismith S, Teixeira-Pinto A, Maze M, Pearce RA, Lennertz R, Sanders RD. Resolution of elevated interleukin-6 after surgery is associated with return of normal cognitive function. Br J Anaesth. 2023 Oct;131(4):694-704. doi: 10.1016/j.bja.2023.05.023. Epub 2023 Jun 27. PMID 37385855
- [Derived] Payne T, Taylor J, Casey C, Kunkel D, Parker M, Blennow K, Zetterberg H, Pearce RA, Lennertz RC, Sanders RD. Prospective analysis of plasma amyloid beta and postoperative delirium in the Interventions for Postoperative Delirium: Biomarker-3 study. Br J Anaesth. 2023 May;130(5):546-556. doi: 10.1016/j.bja.2023.01.020. Epub 2023 Feb 25. PMID 36842841
- [Derived] Taylor J, Payne T, Casey C, Kunkel D, Parker M, Rivera C, Zetterberg H, Blennow K, Pearce RA, Lennertz RC, McCulloch T, Gaskell A, Sanders RD. Sevoflurane dose and postoperative delirium: a prospective cohort analysis. Br J Anaesth. 2023 Feb;130(2):e289-e297. doi: 10.1016/j.bja.2022.08.022. Epub 2022 Oct 1. PMID 36192219
- [Derived] Taylor J, Parker M, Casey CP, Tanabe S, Kunkel D, Rivera C, Zetterberg H, Blennow K, Pearce RA, Lennertz RC, Sanders RD. Postoperative delirium and changes in the blood-brain barrier, neuroinflammation, and cerebrospinal fluid lactate: a prospective cohort study. Br J Anaesth. 2022 Aug;129(2):219-230. doi: 10.1016/j.bja.2022.01.005. Epub 2022 Feb 8. PMID 35144802
- [Derived] Tanabe S, Parker M, Lennertz R, Pearce RA, Banks MI, Sanders RD. Reduced Electroencephalogram Complexity in Postoperative Delirium. J Gerontol A Biol Sci Med Sci. 2022 Mar 3;77(3):502-506. doi: 10.1093/gerona/glab352. PMID 34958346
- [Derived] White MF, Tanabe S, Casey C, Parker M, Bo A, Kunkel D, Nair V, Pearce RA, Lennertz R, Prabhakaran V, Lindroth H, Sanders RD. Relationships between preoperative cortical thickness, postoperative electroencephalogram slowing, and postoperative delirium. Br J Anaesth. 2021 Aug;127(2):236-244. doi: 10.1016/j.bja.2021.02.028. Epub 2021 Apr 15. PMID 33865555
- [Derived] Ballweg T, White M, Parker M, Casey C, Bo A, Farahbakhsh Z, Kayser A, Blair A, Lindroth H, Pearce RA, Blennow K, Zetterberg H, Lennertz R, Sanders RD. Association between plasma tau and postoperative delirium incidence and severity: a prospective observational study. Br J Anaesth. 2021 Feb;126(2):458-466. doi: 10.1016/j.bja.2020.08.061. Epub 2020 Nov 20. PMID 33228978
- [Derived] Tanabe S, Mohanty R, Lindroth H, Casey C, Ballweg T, Farahbakhsh Z, Krause B, Prabhakaran V, Banks MI, Sanders RD. Cohort study into the neural correlates of postoperative delirium: the role of connectivity and slow-wave activity. Br J Anaesth. 2020 Jul;125(1):55-66. doi: 10.1016/j.bja.2020.02.027. Epub 2020 Jun 1. PMID 32499013